CLINICAL TRIAL: NCT02464371
Title: Interest of Plasma microRNAs Assay in ICU Acquired Muscle Weakness Diagnosis
Brief Title: Interest of Plasma microRNAs
Acronym: µARN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1508014
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Septic Shock
Keywords: muscle weakness; microRNAs; septic shock
MeSH Terms: conditions — Shock, Septic; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn to compare the kinetics of microRNAs (miR-1, miR-21, miR-133, miR-155, miR-206, miR-208a, miR-208b, miR-486, miR-499).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU acquired muscle weakness (IAMW) group +: The Medical Research Council score (MRC score) is lower than 48, defining an ICU acquired muscle weakness (IAMW).
  Kinetic of microRNAs is measured
  Interventions: Other: kinetic of microRNAs
- ICU acquired muscle weakness (IAMW) group -: The Medical Research Council score (MRC score) is higher than 48. Kinetic of microRNAs is measured
  Interventions: Other: kinetic of microRNAs

INTERVENTIONS:
Other: kinetic of microRNAs — blood samples will be drawn to measure microRNAs

SUMMARY:
ICU acquired muscle weakness (IAMW) is a common disease that is associated with high morbidity and mortality. Patients with septic shock are particularly at risk.

The diagnosis of IAMW is clinical and based on the rating of the Medical Research Council score (MRC score). A MRC score lower than 48 defines the IAMW. But this evaluation is only usable in sufficiently awaken patients.

Several studies have highlighted the role of microRNAs in regulating physiological processes and diseases related to the skeletal muscles. To date, no study was interested in IAMW.

The aim of this study is to compare the microRNA detection kinetics on the appearance of IAMW.

In septic shock patients, the kinetics of nine microRNAs will be compared between two groups: those with IAMW (IAMW + group) and those without IAMW (IAMW - group).

DETAILED DESCRIPTION:
MicroRNAs (miR-1, miR-21, miR-133, miR-155, miR-206, miR-208a, miR-208b, miR-486, miR-499) will be measured at day 1, day 2, day 5 and day 7 after septic shock onset.

ELIGIBILITY:
Inclusion Criteria:

Patients with septic shock criteria:

* At least two of the following criteria: temperature < 36 ° C or > 38 ° C, heart rate > 90 beats / minute, respiratory rate> 20 breaths / minute or PaCO2 < 32mmHg, leukocytes > 12,000 / mm3 or < 4000 / mm3
* Refractory Hypotension (blood pressure < 90mmHg or need norepinephrine) or lactate ≥ 4 mmol / L

Exclusion Criteria:

* Age<18years
* Patients with preexisting neuromuscular disease
* Pregnancy
* Moribund patients with early therapeutic limitation
* Patients who had a seizure in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: septic shock patients admitted into ICU.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-13 (Actual)

PRIMARY OUTCOMES:
Values of microRNAs between day 1 and day 7 | Day 7
  Values of microRNAs measured between day 1 and day 7 in the 2 groups (IAMW+ group and IAMW- group).

SECONDARY OUTCOMES:
predictive threshold of evolution to the IAMW | Day 1
  From the values of each microRNAs measured at D1, D3, D5 and D7, a predictive threshold of evolution to the IAMW will be sought by the analysis of a ROC curve. The kinetics of microRNAs will be compared between survivors and non-survivors at the discharge.
predictive threshold of evolution to the IAMW | Day 3
  From the values of each microRNAs measured at D1, D3, D5 and D7, a predictive threshold of evolution to the IAMW will be sought by the analysis of a ROC curve. The kinetics of microRNAs will be compared between survivors and non-survivors at the discharge.
predictive threshold of evolution to the IAMW | Day 5
  From the values of each microRNAs measured at D1, D3, D5 and D7, a predictive threshold of evolution to the IAMW will be sought by the analysis of a ROC curve. The kinetics of microRNAs will be compared between survivors and non-survivors at the discharge.
predictive threshold of evolution to the IAMW | Day 7
  From the values of each microRNAs measured at D1, D3, D5 and D7, a predictive threshold of evolution to the IAMW will be sought by the analysis of a ROC curve. The kinetics of microRNAs will be compared between survivors and non-survivors at the discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome MOREL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Ch Roanne, Roanne
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No